CLINICAL TRIAL: NCT04458428
Title: The Role of Postoperative SMS Based Patient Education in Spine Patients
Brief Title: Short Message Service Based Patient Education in Spine Patients
Acronym: SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Ryan Spiker, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 98177
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Patient Satisfaction
Keywords: Spine Surgery; Short Message Service (SMS); Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No other non-standard of care activities will be performed
- Intervention (Experimental): Will be signed up for the automated short message service (SMS)
  Interventions: Other: SMS

INTERVENTIONS:
Other: SMS — Patients who are randomized to the intervention arm will be signed up for the automated SMS program. This cohort will receive text messages after surgery, timed from the day of discharge through 14 days post-op. Patients in this cohort will receive text messages each day. The number of text messages varies on patient interest and "yes" responses to see additional information.
  Arms: Intervention

SUMMARY:
The investigators primary objective is to evaluate whether an SMS based patient education program improves patient satisfaction.

DETAILED DESCRIPTION:
Back and neck related complaints effect as much as 11% of the U.S. population and are one of the most common presenting complaints at health care visits. A small subset of these patients receive spine surgery of various types in the hopes of alleviating symptoms that are recalcitrant to conservative management. The utilization of spine surgery has been rapidly increasing.2 An estimated 413,000 spinal fusions were performed in the U.S. in 2008 accounting for almost $34 billion in charges.

Patient satisfaction has become an increasingly important measure of healthcare quality. This paradigm shift is evident in the changing reimbursement models used by the Centers for Medicare and Medicaid Services (CMS). Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) is a survey-based assessment of patient satisfaction that was initially developed in 2002. Currently, HCAHPS provides the ability to compare patient satisfaction with the care they receive at various healthcare systems across the country. These scores are used as part of a value-based purchasing initiative that can lead to a hospital gaining or losing as much as 1.5% of their annual medicare revenue as a result of patient satisfaction based incentives. This presents an important opportunity to optimize patient satisfaction in order to both improve patient care and preserve hospital income.

A number of novel text-message based applications have been developed for healthcare use in various settings. In the surgical setting text messaging has been used to provide pre-operative education modules, as well as to track medication adherence after transplant. This study aims to develop and critically evaluate, a text-messaging based patient education system aimed at improving patient satisfaction with the post-operative course after spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and over undergoing spine surgery at the University of Utah

Exclusion Criteria:

* Patients under 18 years of age.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
SpineFriend Postoperative Questionnaire | Follow Up Visits at 2 or 6 weeks
  Patient satisfaction will consist of the SpineFriend Postoperative Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Spiker, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States